CLINICAL TRIAL: NCT00837538
Title: A Comparison of Spinal Mouse® and X-ray Film to Measure a Instability of Lumbar Spine
Brief Title: Screening of Instability of the Spinal Column With Spinal Mouse® and X-ray
Status: Completed | Type: Observational
Sponsor: Jyväskylä Central Hospital (Other)
Responsible Party: Ylinen Jari, MD, PhD, Jyväskylä Central Hospital
Other Study IDs: KSSHP 63/2007; KSSHP 63/2007
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Last update posted 2011-03-21 (Estimated); Status verified 2011-03

CONDITIONS: Instability of Lumbar Spine
Keywords: Spinal sagittal range of motion; Intersegmental range of motion; Spinal Mouse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Back pain: Persons with back pain and supposed instability of lumbar spine

SUMMARY:
The SpinalMouse is a computer-assisted medical device that measures and graphically reports on posture and range of motion of the axial spine. The data has shown to be highly valid and reproducible while compared to x-ray film. The aim of the study is to evaluate if the Spinal Mouse is a reliable clinical diagnostic device to screen those patients having instability in the lumbar area.

ELIGIBILITY:
Inclusion Criteria:

* supposed instability of lumbar spine

Exclusion Criteria:

* not willing to participate to study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: persons of Central finland Health Care District
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Sagittal spinal range of motion | One measurement before or after x-ray film

SECONDARY OUTCOMES:
Pain; pain drawing, VAS | Once in the same day with range of motion measurements
Oswestry Disability Questionnaire | Once in the same day with range of motion measurements
Questionnaire; socio-demographic variables, back/leg trouble history | Once in the same day with range of motion measurements

CONTACTS AND LOCATIONS:
Overall Officials: Jari Ylinen, MD, Phd, Study Director — Central Finland Health Care District; Mirja Vuorenmaa, M.Sc., Principal Investigator — Central Finland Heallth Care District; Kirsi Piitulainen, M. Sc., Principal Investigator — Central Finland Care District; Arja Häkkinen, Study Chair — Central Finland Heallth Care District, University of Jyväskylä
Locations (1):
- Central Finland Health Care District, Jyväskylä, Finland